CLINICAL TRIAL: NCT02002117
Title: Genotyping of Non-small Cell Lung Cancer Cells - A Study of Taiwan Lung Cancer Clinical Trial Consortium (TALCC)
Brief Title: Genotyping of Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201103039RB
Record Dates: First submitted 2013-09-09; First posted 2013-12-05 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Non-small Cell Lung Cancer; Gene Abnormality
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — tissue and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DNA mass spectrometry: DNA mass spectrometry
  Interventions: Other: DNA mass

INTERVENTIONS:
Other: DNA mass — DNA mass spectrometry

SUMMARY:
The logical next step is to integrate molecular profiling into the care of all patients with NSCLC.

DETAILED DESCRIPTION:
NSCLC is an area of oncology in which clinicians are beginning to use specific tumor-associated molecular aberrations to assign and/or prioritize targeted therapies for patients. At this early stage, multiple hurdles remain before molecular profiling becomes a routine part of thoracic oncology practice. In particular, to develop specific targeted therapies for patients whose tumors harbor rare mutations, it will be important to identify appropriate candidates, design the appropriate trials, and execute the trials with adequate numbers to achieve the necessary endpoints. Implementation will facilitate realization of the promise of molecularly tailored therapy, which could lead to more effective treatments with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have participated or will be participating a lung cancer clinical trial that use EGFR-TKI or chemotherapy as first line or second line treatment.
2. Pathologic or cytological confirmation of non-small cell lung cancer (NSCLC) with available tissue
3. Patients must understand and provide written informed consent prior to initiation of any study-specific procedures
4. Have a life expectancy 3 months.
5. Have stage IV NSCLC (AJCC, 7th Edition)
6. No or one prior systemic therapy for advanced or metastatic NSCLC 6.1.Adjuvant chemotherapy: The adjuvant chemotherapy (e.g. vinorelbine / cisplatin) should be counted as one prior systemic therapy if the interval between the completion of adjuvant chemotherapy and the documentation of recurrence within 12 months.

   6.2.Maintenance therapy: The maintenance therapy (e.g. pemetrexed) following the first-line systemic chemotherapy which achieved complete response, partial response, or stable disease should not be counted as one prior systemic therapy if the maintenance drug was used in first-line combination therapy
7. ≥20 years
8. ECOG performance status 0 - 2
9. If there is no available archived tissue, the subject must consent to undergo a biopsy or surgical procedure to obtain tissue within 1 month prior to study entry, which may or may not be part of the patient's routine care for their malignancy.

Exclusion Criteria:

1. Prior history of another malignancy (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study entry.
2. Known HIV infection.
3. If subject has no archival tissue and refuse to do any biopsy or surgery for molecular testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to collect 300 EGFR mutation positive samples (approximately 200 de novo, 100 after treatment), 200 EGFR wild type adenocarcinoma patients and 100 other NSCLC patients in 3 years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
frequency of individual genotyping | 2 months
  To determine the frequency of individual genotyping in cancer cells of advanced non-small cell lung cancer (NSCLC) patients who have participated or will commence the clinical trial.

SECONDARY OUTCOMES:
determine the frequency by DNA mass spectrometry | 2 months
  To determine the frequency with which molecular profiling of a NSCLC patient's tumor by DNA mass spectrometry yields a target against which there is approved or investigational therapeutic regimen.
response rate | 1 year
  To determine the response rate according to RECIST, progression-free, and overall survival in patients with advanced NSCLC whose therapy is selected by molecular profile.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, PhD, Principal Investigator
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan